CLINICAL TRIAL: NCT06061107
Title: Effects of Intervention on Hope, Anxiety, and Attitudes and Behavioral Intentions of Advance Care Planning in Older Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202308006RINC
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2023-09

CONDITIONS: Advance Care Planning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handbook for Geriatric Prearranged Medical Care Consultation (Experimental): The experimental group utilized a cartoon version of the "Advance Care Consultation for the Elderly" manual to facilitate the ACP process, which encompassed three components: an introduction to ACP, an overview of terminal medical care, and a discussion about the participants' preferences for their past, current, and future required medical care.
  Interventions: Behavioral: The cartoon version of the "ACP for Seniors" brochure
- Control group (No Intervention): No Intervention: standard clinical care

INTERVENTIONS:
Behavioral: The cartoon version of the "ACP for Seniors" brochure — The experimental group utilized a cartoon version of the "Advance Care Consultation for the Elderly" manual to facilitate the ACP process, which encompassed three components: an introduction to ACP, an overview of terminal medical care, and a discussion about the participants' preferences for their past, current, and future required medical care. There are three measurement time points: pre-test, two weeks after intervention, and one month after intervention.
  Arms: Handbook for Geriatric Prearranged Medical Care Consultation

SUMMARY:
The study aims to explore the impact of advance care planning on the attitudes, behavioral intentions, hopes, and anxiety of elderly people with cancer on advance care planning with the assistance of the "Advance Care Consultation for the Elderly" manual.

DETAILED DESCRIPTION:
The experimental group used the cartoon version of the "Advance Care Consultation for the Elderly" manual to guide the ACP process. The process included three parts: an introduction to ACP, an introduction to terminal medical care, and a discussion of what the participants wanted to do about their own health in the past, present, and future required medical care. The estimated time to lead and conduct the ACP conversation is approximately 40 minutes. The control group maintained routine care. The measurement tools are the Advance Care Planning Attitude Scale, Behavioral Intention Scale, Chinese version of Situational Anxiety Inventory-Situational Anxiety Inventory (STAI-S), and Hope State Inventory (Herth Hope Index, HHI) ). There are three measurement time points: pre-test, two weeks after intervention, and one month after intervention. Expected research results: It is expected that intervention measures can improve the positive attitudes and behavioral intentions of elderly people with cancer towards ACP while maintaining their sense of hope without increasing anxiety. It is hoped that the intervention of ACP can enhance the exploration of their own medical preferences and values by the elderly with cancer, and help them become more aware of their own choices and needs when facing treatment decisions in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients aged 65 years or older.
2. Patients currently undergoing cancer treatment.
3. Clear consciousness and able to communicate in Mandarin or Taiwanese.
4. Score of 8 points or higher (inclusive) on the Short Portable Mental State Questionnaire (SPMSQ).

Exclusion Criteria:

1. Individuals with a score of 7 points or lower (inclusive) on the Short Portable Mental State Questionnaire (SPMSQ).
2. Individuals who have not been informed about their cancer diagnosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Attitude Scale | three measurement time points: pre-test, two weeks after intervention, and one month after intervention.
  The questionnaire is scored using a 5-point Likert scale. There are a total of 12 questions, resulting in a total score ranging from 24 to 120, with responses ranging from "strongly disagree" (1 point) to "strongly agree" (5 points) . A higher score indicates a more positive attitude among the elderly towards advance care planning.
Behavioral Intention Scale | three measurement time points: pre-test, two weeks after intervention, and one month after intervention.
  The scale is scored using a 5-point Likert scale. There are a total of six questions, resulting in a total score ranging from 6 to 30, with responses ranging from "very unlikely" (1 point) to "very likely" (5 points)
State Anxiety, A-State，STAI-S | three measurement time points: pre-test, two weeks after intervention, and one month after intervention.
  The scale consists of 20 questions, each with 4 options: "completely does not fit," "fits slightly," "fits," and "fits very well." Out of these, 10 questions are positively framed (3, 4, 6, 7, 9, 12, 13, 14, 17, and 18). The scoring is as follows: "1 point" for "completely does not fit," "2 points" for "fits slightly," "3 points" for "fits," and "4 points" for "fits very well." The remaining ten questions are negatively framed, and scoring is reversed, with "4 points" for "completely does not fit," "3 points" for "fits slightly," "2 points" for "fits," and "1 point" for "fits very well." The total score ranges from 20 to 80 points. A higher score indicates a higher level of anxiety, with scores of 20 to 39 indicating mild anxiety, 40 to 59 indicating moderate anxiety, and 60 to 80 indicating severe anxiety.
Herth Hope Index, HHI | three measurement time points: pre-test, two weeks after intervention, and one month after intervention.
  The scale is scored using a 4-point Likert scale, with "1 point" indicating "strongly disagree" and "4 points" indicating "strongly agree," resulting in a total score ranging from 12 to 48 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hsu Ya Hui, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu YH, Wang MH, Hu WY, Ke LS. Effects of advance care planning on hope, anxiety, attitudes, and behavioral intentions in older adults with cancer: A randomized controlled study. Support Care Cancer. 2025 Aug 30;33(9):822. doi: 10.1007/s00520-025-09866-z. PMID 40884542